CLINICAL TRIAL: NCT01702805
Title: Transfusion of Prematures (TOP) Trial: Does a Liberal Red Blood Cell Transfusion Strategy Improve Neurologically-Intact Survival of Extremely-Low-Birth-Weight Infants as Compared to a Restrictive Strategy?
Brief Title: Transfusion of Prematures Trial
Acronym: TOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NICHD-NRN-0050; U01HL112776 (NIH); U01HL112748 (NIH)
Record Dates: First submitted 2012-08-30; First posted 2012-10-08 (Estimated); Results first posted 2022-02-11 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Infant, Newborn, Diseases; Infant, Extremely Low Birth Weight; Infant, Small for Gestational Age; Bronchopulmonary Dysplasia (BPD); Anemia
Keywords: NICHD Neonatal Research Network; Very Low Birth Weight (VLBW); Extremely Low Birth Weight (ELBW); Transfusions
MeSH Terms: conditions — Infant, Newborn, Diseases; Bronchopulmonary Dysplasia; Anemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low Threshold Transfusion (Active Comparator): Transfusions will be administered using a lower threshold hemoglobin value. The low threshold values reflect more common practice, so this is considered the 'usual treatment' group
  Interventions: Procedure: Restricted red cell transfusion
- High Threshold Transfusion (Active Comparator): Transfusions will be administered using a higher threshold hemoglobin value.
  Interventions: Procedure: Liberal Cell Transfusion

INTERVENTIONS:
Procedure: Liberal Cell Transfusion
  Arms: High Threshold Transfusion
Procedure: Restricted red cell transfusion
  Arms: Low Threshold Transfusion

SUMMARY:
The objective of the TOP trial is to determine whether higher hemoglobin thresholds for transfusing ELBW infants resulting in higher hemoglobin levels lead to improvement in the primary outcome of survival and rates of neurodevelopmental impairment (NDI) at 22-26 months of age, using standardized assessments by Bayley.

DETAILED DESCRIPTION:
Long-term outcomes of extremely low birth weight (ELBW) preterm infants, those weighing less than or equal to 1000 g at birth, are poor and pose a major health care burden. Virtually all of these infants are transfused, but at inconsistent hemoglobin (Hgb) thresholds.

The investigators propose in TOP to randomize infants less than or equal to 1000 g BW and gestational age at least 22 weeks but less than 29 weeks to receive red blood cell (RBC) transfusions according to one of two strategies of Hgb thresholds, either a high Hgb (liberal transfusion) or a low Hgb (restrictive transfusion) algorithm. It is currently unknown which transfusion strategy is superior. TOP is powered to demonstrate which strategy reduces the primary outcome of death or neurodisability in survivors at 22-26 months.

A secondary study entitled "Effect of Blood Transfusion Practices on Cerebral and Somatic Oximetry", also known as the NIRS study, will determine differences in cerebral oxygenation and fractional tissue oxygen extraction with NIRS between high and low hemoglobin threshold groups during red blood cell transfusions. The investigators also propose to determine whether abnormal cerebral NIRS measures are a better predictor of NDI than hemoglobin alone and whether abnormal mesenteric NIRS measures are associated with the development of NEC within the 48 hours following a transfusion.

A secondary study entitled "Economic Evaluation Ancillary to the Transfusion of Prematures Randomized Controlled Trial" will determine whether higher transfusion threshold will result in lower total costs to society over the first 22 to 26 corrected months of life and estimate the incremental cost-effectiveness ratio for survival without neurodevelopmental impairment, from the perspective of society, the third-party payer, and the family.

Extended follow-up: Subjects will be seen for a follow-up visit at 5-6 years corrected age to assess neurological and functional outcomes at early school age based on neonatal transfusion threshold.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight less than or equal to 1000 grams.
* Gestational age at least 22 weeks but less than 29 weeks
* Admitted to the NICU within 48 hours of life

Exclusion Criteria:

* Considered nonviable by the attending neonatologist
* Cyanotic congenital heart disease
* Parents opposed to the transfusion of blood
* Parents with hemoglobinopathy or congenital anemia
* In-utero fetal transfusion
* Twin-to-twin transfusion syndrome
* Isoimmune hemolytic disease
* Lack of parental consent
* Severe acute hemorrhage, acute shock, sepsis with coagulopathy, or need for perioperative transfusion.
* Prior blood transfusion on clinical grounds beyond the first 6 hours of life
* Infant has received erythropoietin prior to randomization, or is intended to receive erythropoietin through the neonatal course
* Congenital condition, other than premature birth, that adversely affects life expectancy or neurodevelopment.
* High probability that the family is socially disorganized to the point of being unable to attend follow-up at 22-26 months.

Max Age: 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1824 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2025-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele C Walsh, MD, Principal Investigator — Case Western Reserve University, Rainbow Babies and Children's Hospital; Abhik Das, PhD, Principal Investigator — RTI International; Beena Sood, MD, Principal Investigator — Wayne State University; Abbot R Laptook, MD, Principal Investigator — Brown University, Women & Infants Hospital of Rhode Island; Michael Cotten, MD, Principal Investigator — Duke University; Ravi Patel, MD, Principal Investigator — Emory University; Greg Sokol, MD, Principal Investigator — Indiana University; Krisa P Van Meurs, MD, Principal Investigator — Stanford University; Brenda Poindexter, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Waldemar A Carlo, MD, Principal Investigator — University of Alabama at Birmingham; Kristi L Watterberg, MD, Principal Investigator — University of New Mexico; Myra Wyckoff, MD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas; Kathleen A Kennedy, MD, MPH, Principal Investigator — The University of Texas Health Science Center, Houston; Carl T D'Angio, MD, Principal Investigator — University of Rochester; Pablo Sanchez, MD, Principal Investigator — Research Institute at Nationwide Children's Hospital; William Truog, MD, Principal Investigator — Children's Mercy Hospital Kansas City; Uday Devaskar, MD, Principal Investigator — University of California, Los Angeles; Haresh M Kirpalani, MD, Study Director — University of Pennsylvania; Bradley Yoder, MD, Principal Investigator — University of Utah
Locations (20):
- United States (20):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California - Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Wayne State University, Detroit, Michigan
  - Children's Mercy Hospital, Kansas City, Missouri
  - University of New Mexico, Albuquerque, New Mexico
  - University of Rochester, Rochester, New York
  - RTI International, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Research Institute at Nationwide Children's Hospital, Columbus, Ohio
  - Univeristy of Pennsylvania, Philadelphia, Pennsylvania
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
NIH has had a long-standing policy to share and make available to the public the results and accomplishments of the activities that it funds. The NRN plans to share de-identified data after final publication in an NIH supported data repository such as the NICHD Data and Specimen Hub (https://dash.nichd.nih.gov)

REFERENCES:
- [Derived] Conrad AL, DeMauro SB, Kirpalani H, Ziolkowski K, Hintz SR, Vohr BR, Watson V, Colaizy TT, Bell EF, Brumbaugh JE, Bann CM, Tan SM, Newman JE, Das A. The transfusion of prematures early school age follow-up (TOP 5): protocol for a longitudinal cohort study. BMC Pediatr. 2025 May 15;25(1):387. doi: 10.1186/s12887-025-05732-3. PMID 40375228
- [Derived] Salas AA, Gunn E, Carlo WA, Bell EF, Das A, Josephson CD, Patel RM, Tan S, Kirpalani H; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Neonatal Research Network. Timing of Red Blood Cell Transfusions and Occurrence of Necrotizing Enterocolitis: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2024 May 1;7(5):e249643. doi: 10.1001/jamanetworkopen.2024.9643. PMID 38700862
- [Derived] Chock VY, Kirpalani H, Bell EF, Tan S, Hintz SR, Ball MB, Smith E, Das A, Loggins YC, Sood BG, Chalak LF, Wyckoff MH, Kicklighter SD, Kennedy KA, Patel RM, Carlo WA, Johnson KJ, Watterberg KL, Sanchez PJ, Laptook AR, Seabrook RB, Cotten CM, Mancini T, Sokol GM, Ohls RK, Hibbs AM, Poindexter BB, Reynolds AM, DeMauro SB, Chawla S, Baserga M, Walsh MC, Higgins RD, Van Meurs KP; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Tissue Oxygenation Changes After Transfusion and Outcomes in Preterm Infants: A Secondary Near-Infrared Spectroscopy Study of the Transfusion of Prematures Randomized Clinical Trial (TOP NIRS). JAMA Netw Open. 2023 Sep 5;6(9):e2334889. doi: 10.1001/jamanetworkopen.2023.34889. PMID 37733345
- [Derived] Kirpalani H, Bell EF, Hintz SR, Tan S, Schmidt B, Chaudhary AS, Johnson KJ, Crawford MM, Newman JE, Vohr BR, Carlo WA, D'Angio CT, Kennedy KA, Ohls RK, Poindexter BB, Schibler K, Whyte RK, Widness JA, Zupancic JAF, Wyckoff MH, Truog WE, Walsh MC, Chock VY, Laptook AR, Sokol GM, Yoder BA, Patel RM, Cotten CM, Carmen MF, Devaskar U, Chawla S, Seabrook R, Higgins RD, Das A; Eunice Kennedy Shriver NICHD Neonatal Research Network. Higher or Lower Hemoglobin Transfusion Thresholds for Preterm Infants. N Engl J Med. 2020 Dec 31;383(27):2639-2651. doi: 10.1056/NEJMoa2020248. PMID 33382931
- See also: NICHD NRN Website — http://neonatal.rti.org/
- See also: NICHD Pregnancy & Perinatology Branch — https://www.nichd.nih.gov/about/org/der/branches/ppb

RESULTS

PARTICIPANT FLOW:
Groups:
- High Tranfusion Threshold: Transfusions were administered using a higher threshold hemoglobin value. AKA "Liberal Cell Transfusion" group.
- Low Transfusion Threshold: Transfusions were administered using a lower threshold hemoglobin value. The low threshold values reflect more common practice, so this is considered the 'usual treatment' group. AKA "Restricted Red Cell Transfusion" group.
Period: Overall Study
Arm/Group | High Tranfusion Threshold | Low Transfusion Threshold
Started | 911 | 913
Completed Assessment for Neurodevelopmental Impairment | 699 | 712
Died After Discharge | 19 | 10
Died Before Discharge | 127 | 125
Survived to Discharge | 781 | 781
Completed (Complete data for Primary Outcome, Death or Neurodevelopmental Impairment) | 845 | 847
Not Completed | 66 | 66
Not completed — Data withdrawn prior to hospital discharge | 3 | 7
Not completed — Incomplete Follow-up | 18 | 15
Not completed — Vital Status Assessment Only | 40 | 39
Not completed — Lost to Follow-up | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- High Transfusion Threshold: Transfusions were administered using a higher threshold hemoglobin value. AKA 'Liberal Cell Transfusion' group.
- Low Transfusion Threshold: Transfusions were administered using a lower threshold hemoglobin value. The low threshold values reflect more common practice, so this is considered the 'usual treatment' group. AKA 'Restricted Red C
- Total: Total of all reporting groups
Arm/Group | High Transfusion Threshold | Low Transfusion Threshold | Total
Number analyzed (Participants) | 911 | 913 | 1824
Age, Continuous [Mean (Standard Deviation); unit: weeks] — Age refers to the infant and is measured as gestational age in weeks
  weeks | 25.9 (1.5) | 25.9 (1.5) | 25.9 (1.5)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 488 | 462 | 950
  Male | 423 | 451 | 874
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 149 | 150 | 299
  Not Hispanic or Latino | 754 | 753 | 1507
  Unknown or Not Reported | 8 | 10 | 18
Maternal Race, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 6 | 14
  Asian, Native Hawaiian, or Other Pacific Islander | 25 | 35 | 60
  Black or African American | 423 | 395 | 818
  More Than One Race | 20 | 15 | 35
  Unknown or Not Reported | 16 | 25 | 41
  White | 419 | 437 | 856

OUTCOME MEASURES:

1. Primary Outcome: Death or Neurodevelopmental Impairment
Description: A composite outcome that measures the occurrence of death or neurodevelomental impairment between birth and 22-26 months corrected age.
Time Frame: Birth to 22-26 months corrected age
Population: The analysis population includes all randomized infants with available data for death and/or neurodevelopmental impairment.
Measure: Count of Participants; unit: Participants
Arm/Group | High Transfusion Threshold | Low Transfusion Threshold
Number analyzed (Participants) | 845 | 847
Participants
  Death or Neurodevelopmental Impairment | 423 | 422
  No Death nor Neurodevelopmental Impairment | 422 | 425
Statistical Analysis 1: Comparison: Low Transfusion Threshold; Null hypothesis: A higher hemoglobin threshold for red-cell transfusions, as compared with a lower threshold, will not reduce nor increase the incidence of death or neurodevelopmental impairment in infants at 22 to 26 months of age corrected for prematurity; Test type: Superiority; p = 0.93, Robust Poisson Regression; The relative risk was adjusted for birth-weight and center stratum; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.92 to 1.10]

2. Primary Outcome: Death
Description: This is measured as Yes if an infant died between birth and 22-26 months corrected age; Otherwise, No.
Time Frame: Birth to 22-26 months corrected age
Population: The analysis population includes all randomized infants with available vital status.
Measure: Count of Participants; unit: Participants
Arm/Group | High Transfusion Threshold | Low Transfusion Threshold
Number analyzed (Participants) | 903 | 901
Participants
  Death | 146 | 135
  No Death | 757 | 766

3. Primary Outcome: Neurodevelopmental Impairment
Description: This is measured as Yes if any hearing impairment or visual impairment is noted, if severe or moderate cerebral palsy is noted, or if the cognitive score of the Bayley III score is more than 1 standard deviation below the average; Otherwise, No.
Time Frame: at 22-26 months corrected age
Population: The analysis population includes all randomized infants with available data for neurodevelopmental impairment.
Measure: Count of Participants; unit: Participants
Arm/Group | High Transfusion Threshold | Low Transfusion Threshold
Number analyzed (Participants) | 699 | 712
Participants
  Neurodevelopmental Impairment | 277 | 287
  No Neurodevelopmental Impairment | 422 | 425

4. Primary Outcome: Cognitive Delay
Description: This is measured as Yes if the Bayley Scale of Infant and Toddler Development (BSID)-III cognitive score is more than 1 standard deviation below the average; Otherwise, No.
Time Frame: at 22-26 months corrected age
Population: The analysis population includes all randomized infants with available data at the two-year followup.
Measure: Count of Participants; unit: Participants
Arm/Group | High Transfusion Threshold | Low Transfusion Threshold
Number analyzed (Participants) | 695 | 712
Participants
  Cognitive Delay | 269 | 270
  No Cognitive Delay | 426 | 442

5. Primary Outcome: Moderate or Severe Cerebral Palsy
Description: This is measured as Yes if the Gross Motor Function Classification System (GMFCS) score is level II or higher; Otherwise, No. Higher values of the GMFCS are worse than lower values; a level of "I" denotes mild cerebral palsy (CP); level "II" or "III" moderate CP; level "IV" or "V" severe CP.
Time Frame: at 22-26 months corrected age
Population: The analysis population includes all randomized infants with available data at the two-year followup.
Measure: Count of Participants; unit: Participants
Arm/Group | High Transfusion Threshold | Low Transfusion Threshold
Number analyzed (Participants) | 711 | 720
Participants
  Moderate or Severe Cerebral Palsy | 48 | 55
  Mild or No Cerebral Palsy | 663 | 665

6. Primary Outcome: Severe Vision Impairment
Description: This is measured as Yes if the corrected visual acuity in the better eye of less than 20/200; Otherwise, No.
Time Frame: at 22-26 months corrected age
Population: The analysis population includes all randomized infants with available data at the two-year followup.
Measure: Count of Participants; unit: Participants
Arm/Group | High Transfusion Threshold | Low Transfusion Threshold
Number analyzed (Participants) | 713 | 720
Participants
  No Severe Vision Impairment | 708 | 714
  Severe Vision Impairment | 5 | 6

7. Primary Outcome: Severe Hearing Impairment
Description: This is measured as Yes if bilateral hearing loss occurred for which hearing aids or cochlear implants were warranted; Otherwise, No.
Time Frame: at 22-26 months corrected age
Population: The analysis population includes all randomized infants with available data at the two-year followup.
Measure: Count of Participants; unit: Participants
Arm/Group | High Transfusion Threshold | Low Transfusion Threshold
Number analyzed (Participants) | 710 | 715
Participants
  No Severe Hearing Impairment | 696 | 690
  Severe Hearing Impairment | 14 | 25

8. Secondary Outcome: Survival to Discharge Without Severe Complications
Description: This is measured as Yes if survived to discharge without severe morbidity, defined as bronchopulmonary dysplasia, retinopathy of prematurity (stage 3 or higher or requiring treatment), or serious brain abnormality; Otherwise, No.
Time Frame: Birth to initial hospital discharge or to death if it occurs earlier (a median of 97 days)
Population: The analysis population includes all randomized infants with available data up to hospital discharge or death.
Measure: Count of Participants; unit: Participants
Arm/Group | High Transfusion Threshold | Low Transfusion Threshold
Number analyzed (Participants) | 901 | 888
Participants
  No Survival to Discharge Without Severe Complications | 644 | 614
  Survival to Discharge Without Severe Complications | 257 | 274

9. Secondary Outcome: Bronchopulmonary Dysplasia, Diagnosed on the Basis of the Need for Supplemental Oxygen After a Standardized Oxygen Reduction Test at 36 Weeks of Postmenstrual Age
Description: This is measured as Yes if experienced bronchopulmonary dysplasia, diagnosed on the basis of the need for supplemental oxygen after a standardized oxygen reduction test at 36 weeks of postmenstrual age; Otherwise, No.
Time Frame: at 36 weeks postmenstrual age
Population: The analysis population includes all randomized infants with available data at 36 weeks postmenstrual age.
Measure: Count of Participants; unit: Participants
Arm/Group | High Transfusion Threshold | Low Transfusion Threshold
Number analyzed (Participants) | 795 | 805
Participants
  Bronchopulmonary Dysplasia at 36 Weeks Postmenstrual Age | 469 | 453
  No Bronchopulmonary Dysplasia at 36 Weeks Postmenstrual Age | 326 | 352

10. Secondary Outcome: Retinopathy of Prematurity Stage >=3 or Treatment for That Condition Received
Description: This is measured as Yes if experienced Retinopathy of Prematurity (ROP) Stage >=3 or received treatment for that condition; Otherwise, No. Higher stages of ROP indicate a worse outcome; the stages range from 1 for "mild" disease, to 5 for "severe" disease.
Time Frame: Birth to initial hospital discharge or to death if it occurs earlier (a median of 97 days)
Population: The analysis population includes all randomized infants with available data up to hospital discharge or death.
Measure: Count of Participants; unit: Participants
Arm/Group | High Transfusion Threshold | Low Transfusion Threshold
Number analyzed (Participants) | 797 | 797
Participants
  No Retinopathy of Prematurity at least Stage 3 and did not Receive Treatment for Such Condition | 640 | 660
  Retinopathy of Prematurity at least Stage 3 or Received Treatment for Such Condition | 157 | 137

11. Secondary Outcome: Grade 3 or 4 Intraventricular Hemorrhage, Cystic Periventricular Leukomalacia, or Ventriculomegaly Diagnosed on Ultrasonographic Examination
Description: This is measured as Yes if experienced Grade 3 or 4 intraventricularhemorrhage, cystic periventricular leukomalacia, or ventriculomegaly diagnosed on ultrasonographic examination; Otherwise, No.
Time Frame: Birth to initial hospital discharge or to death if it occurs earlier (a median of 97 days)
Population: The analysis population includes all randomized infants with available data up to hospital discharge or death.
Measure: Count of Participants; unit: Participants
Arm/Group | High Transfusion Threshold | Low Transfusion Threshold
Number analyzed (Participants) | 855 | 859
Participants
  Grade 3 or 4 intraventricular hemorrhage, cystic periventricular leukomalacia, or ventriculomegaly | 146 | 154
  None of the stated head ultrasound diagnoses | 709 | 705

12. Secondary Outcome: Necrotizing Enterocolitis, Bell's Stage >=2
Description: This is measured as Yes if experienced necrotizing enterocolitis (NEC), Bell's stage >=2; Otherwise, No. Higher scores of Bell's staging criteria denote a worse outcome, where "1" denotes suspect, "2" definite and "3" advanced NEC.
Time Frame: Birth to initial hospital discharge or to death if it occurs earlier (a median of 97 days)
Population: The analysis population includes all randomized infants with available data up to hospital discharge or death.
Measure: Count of Participants; unit: Participants
Arm/Group | High Transfusion Threshold | Low Transfusion Threshold
Number analyzed (Participants) | 907 | 906
Participants
  NEC, Bell's Stage >= 2 | 91 | 95
  NEC, Bell's Stage = 1 or no NEC | 816 | 811

13. Secondary Outcome: Number of Transfusions Per Infant
Description: This is measured as the number of protocol compliant transfusions, clinically justified non-protocol transfusions and unjustified non-protocol transfusions (violations)
Time Frame: Birth, up to the earliest of: death, hospital discharge, or 36 weeks postmenstrual age (PMA)
Population: The analysis population includes all randomized infants with available data up to death, hospital discharge, or 36 weeks PMA, whichever occurs first
Measure: Mean (Standard Deviation); unit: Transfusions
Arm/Group | High Transfusion Threshold | Low Transfusion Threshold
Number analyzed (Participants) | 911 | 913
Transfusions | 6.2 (4.3) | 4.4 (4.0)

14. Secondary Outcome: Weight-for-age: Z-score
Description: This is measured as the weight-for-age Z-score at 36 weeks postmenstrual age or at initial hospital discharge, whichever occurs first. The Z-score is determined using Olsen percentile curves, and is derived from a normal distribution, where 0 designates average weight-for-age, and negative scores denote less than average weight-for-age.
Time Frame: at 36 weeks postmenstrual age or initial hospital discharge, whichever occurs first
Population: The analysis population includes all randomized infants with available data at 36 weeks postmenstrual age or at initial hospital discharge, whichever occurs first.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | High Transfusion Threshold | Low Transfusion Threshold
Number analyzed (Participants) | 769 | 774
Z-score | -1.2 (0.8) | -1.3 (0.8)

15. Secondary Outcome: Length-for-age: Z-score
Description: This is measured as the length-for-age Z-score at 36 weeks postmenstrual age or at initial hospital discharge, whichever occurs first. The Z-score is determined using Olsen percentile curves, and is derived from a normal distribution, where 0 designates average length-for-age, and negative scores denote less than average length-for-age.
Time Frame: at 36 weeks postmenstrual age or initial hospital discharge, whichever occurs first
Population: The analysis population includes all randomized infants with available data at 36 weeks postmenstrual age or initial hospital discharge, whichever occurs first.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | High Transfusion Threshold | Low Transfusion Threshold
Number analyzed (Participants) | 715 | 715
Z-score | -1.9 (1.0) | -1.9 (0.9)

16. Secondary Outcome: Head Circumference-for-age: Z-score
Description: This is measured as the head circumference-for-age Z-score at 36 weeks postmenstrual age or at initial hospital discharge, whichever occurs first. The Z-score is determined using Olsen percentile curves, and is derived from a normal distribution, where 0 designates average head circumference-for-age, and negative scores denote less than average head circumference-for-age.
Time Frame: at 36 weeks postmenstrual age or initial hospital discharge, whichever occurs first
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | High Transfusion Threshold | Low Transfusion Threshold
Number analyzed (Participants) | 754 | 766
Z-score | -1.4 (1.0) | -1.4 (1.0)

17. Secondary Outcome: Postmenstrual Age at Final Trachael Extubation
Description: This is measured as the average postmenstrual age (in weeks) at final tracheal extubation in infants who were intubated.
Time Frame: at final trachael extubation, assessed from birth up to the earliest of: death, hospital discharge, or 36 weeks postmenstrual age
Population: The analysis population includes all randomized infants with available data on trachael extubation.
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | High Transfusion Threshold | Low Transfusion Threshold
Number analyzed (Participants) | 796 | 804
Weeks | 30 (3.4) | 30.2 (3.3)

18. Secondary Outcome: Postmenstrual Age at Final Caffeine Dose in Infants Who Received Caffeine Treatment
Description: This is measured as the average postmenstrual age (in weeks) at final caffeine dose in infants who received caffeine treatment.
Time Frame: at final caffeine dose, assessed from birth up to the earliest of: death, hospital discharge, or 36 weeks postmenstrual age
Population: The analysis population includes all randomized infants with available data on caffeine treatment.
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | High Transfusion Threshold | Low Transfusion Threshold
Number analyzed (Participants) | 882 | 887
Weeks | 33.8 (3.0) | 34.0 (2.8)

19. Secondary Outcome: Length of Stay
Description: This is measured as the length of stay (in days) up to initial hospital discharge or death, whichever occurred first.
Time Frame: at initial hospital discharge or at death if it occurs earlier (a median of 97 days)
Population: The analysis population includes all randomized infants with available data up to the initial hospital discharge or death, whichever occurs first.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | High Transfusion Threshold | Low Transfusion Threshold
Number analyzed (Participants) | 908 | 906
Days | 96 [72 to 129] | 97 [75 to 127]

20. Secondary Outcome: Time to Full Enteral Feeding
Description: This is measured as the amount of days it took for full enteral feeding to occur.
Time Frame: at first full enteral feeding, assessed from birth up to initial hospital discharge or to death if it occurs earlier (a median of 97 days)
Population: The analysis population includes all randomized infants with available data on enteral feeding.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | High Transfusion Threshold | Low Transfusion Threshold
Number analyzed (Participants) | 808 | 824
Days | 19.5 [14 to 29] | 19.0 [15 to 30]

21. Secondary Outcome: Severe Cerebral Palsy
Description: This is measured as Yes if Gross Motor Function Classification System (GMFCS) is levels IV or V; Otherwise, No. Higher values of the GMFCS are worse than lower values; a level of "I" denotes mild cerebral palsy (CP); level "II" or "III" moderate CP; level "IV" or "V" severe CP.
Time Frame: at 22-26 months corrected age
Population: The analysis population includes all randomized infants with available data at the two-year followup.
Measure: Count of Participants; unit: Participants
Arm/Group | High Transfusion Threshold | Low Transfusion Threshold
Number analyzed (Participants) | 710 | 720
Participants
  No Severe Cerebral Palsy | 690 | 709
  Severe Cerebral Palsy | 20 | 11

22. Secondary Outcome: Hydrocephalus Shunt
Description: This is measured as Yes if experienced Hydrocephalus shunt by follow-up; Otherwise, No.
Time Frame: Initial hospital discharge to 22-26 months corrected age
Population: The analysis population includes all randomized infants with available data at the two-year followup.
Measure: Count of Participants; unit: Participants
Arm/Group | High Transfusion Threshold | Low Transfusion Threshold
Number analyzed (Participants) | 717 | 728
Participants
  Hydrocephalus Shunt | 20 | 22
  No Hydrocephalus Shunt | 697 | 706

23. Secondary Outcome: Microcephaly
Description: This is measured as a head circumference-for-age Z-score of less than -2; Otherwise, No. The Z-score is determined using WHO percentile curves, and is derived from a normal distribution, where 0 designates average head circumference-for-age, and negative scores denote less than average head circumference-for-age.
Time Frame: at 22-26 months corrected age
Population: The analysis population includes all randomized infants with available data at the two-year followup.
Measure: Count of Participants; unit: Participants
Arm/Group | High Transfusion Threshold | Low Transfusion Threshold
Number analyzed (Participants) | 700 | 710
Participants
  Microcephaly | 61 | 52
  No Microcephaly | 639 | 658

24. Secondary Outcome: Seizure Disorder
Description: This is measured as Yes if experienced one or more seizures since discharge or of regular use of anticonvulsants or seizure medications; Otherwise, No.
Time Frame: Initial hospital discharge to 22-26 months corrected age
Population: The analysis population includes all randomized infants with available data at the two-year followup.
Measure: Count of Participants; unit: Participants
Arm/Group | High Transfusion Threshold | Low Transfusion Threshold
Number analyzed (Participants) | 714 | 726
Participants
  No Seizure disorder | 672 | 685
  Seizure disorder | 42 | 41

25. Secondary Outcome: Respiratory Disease Necessitating Readmission Before Follow-up
Description: This is measured as Yes if obtained Respiratory disease necessitating readmission before follow-up; Otherwise, No.
Time Frame: Initial hospital discharge to 22-26 months corrected age
Population: The analysis population includes all randomized infants with available data at the two-year followup.
Measure: Count of Participants; unit: Participants
Arm/Group | High Transfusion Threshold | Low Transfusion Threshold
Number analyzed (Participants) | 715 | 726
Participants
  No Respiratory disease necessitating readmission before follow-up | 467 | 496
  Respiratory disease necessitating readmission before follow-up | 248 | 230

26. Secondary Outcome: Composite Language Score Less Than 85
Description: This is measured as Yes if scored less than 85 on the Bayley Scale of Infant and Toddler Development (BSID)-III composite language score; Otherwise, No. Higher scores indicate better performance. Composite BSID-III scores of less than 85 are less than 1 standard deviation below the mean of 100.
Time Frame: at 22-26 months corrected age
Population: The analysis population includes all randomized infants with available data at the two-year followup.
Measure: Count of Participants; unit: Participants
Arm/Group | High Transfusion Threshold | Low Transfusion Threshold
Number analyzed (Participants) | 671 | 691
Participants
  Composite language score greater or equal to 85 | 316 | 323
  Composite language score less than 85 | 355 | 368

27. Secondary Outcome: Composite Motor Score Less Than 85
Description: This is measured as Yes if scored less than 85 on the Bayley Scale of Infant and Toddler Development (BSID)-III composite motor score; Otherwise, No. Higher scores indicate better performance. Composite BSID-III scores of less than 85 are less than 1 standard deviation below the mean of 100.
Time Frame: at 22-26 months corrected age
Population: The analysis population includes all randomized infants with available data at the two-year followup.
Measure: Count of Participants; unit: Participants
Arm/Group | High Transfusion Threshold | Low Transfusion Threshold
Number analyzed (Participants) | 678 | 695
Participants
  Composite motor score greater or equal to 85 | 423 | 415
  Composite motor score less than 85 | 255 | 280

28. Secondary Outcome: Composite Cognitive Score Less Than 70
Description: This is measured as Yes if scored less than 85 on the Bayley Scale of Infant and Toddler Development (BSID)-III composite cognitive score; Otherwise, No. Higher scores indicate better performance. Composite BSID-III scores of less than 70 are less than 2 standard deviations below the mean of 100.
Time Frame: at 22-26 months corrected age
Population: The analysis population includes all randomized infants with available data at the two-year followup.
Measure: Count of Participants; unit: Participants
Arm/Group | High Transfusion Threshold | Low Transfusion Threshold
Number analyzed (Participants) | 695 | 712
Participants
  Composite cognitive score greater or equal to 70 | 607 | 616
  Composite cognitive score less than 70 | 88 | 96

29. Secondary Outcome: Composite Language Score Less Than 70
Description: This is measured as Yes if scored less than 85 on the Bayley Scale of Infant and Toddler Development (BSID)-III composite language score; Otherwise, No. Higher scores indicate better performance. Composite BSID-III scores of less than 70 are less than 2 standard deviations below the mean of 100.
Time Frame: at 22-26 months corrected age
Population: The analysis population includes all randomized infants with available data at the two-year followup.
Measure: Count of Participants; unit: Participants
Arm/Group | High Transfusion Threshold | Low Transfusion Threshold
Number analyzed (Participants) | 671 | 691
Participants
  Composite language score greater or equal to 70 | 507 | 528
  Composite language score less than 70 | 164 | 163

30. Secondary Outcome: Composite Motor Score Less Than 70
Description: This is measured as Yes if scored less than 85 on the Bayley Scale of Infant and Toddler Development (BSID)-III composite motor score; Otherwise, No. Higher scores indicate better performance. Composite BSID-III scores of less than 70 are less than 2 standard deviations below the mean of 100.
Time Frame: at 22-26 months corrected age
Population: The analysis population includes all randomized infants with available data at the two-year followup.
Measure: Count of Participants; unit: Participants
Arm/Group | High Transfusion Threshold | Low Transfusion Threshold
Number analyzed (Participants) | 678 | 695
Participants
  Composite motor score greater or equal to 70 | 591 | 596
  Composite motor score less than 70 | 87 | 99

ADVERSE EVENTS:
Time Frame: Birth to 37 weeks PMA
Arm/Group | High Tranfusion Threshold | Low Transfusion Threshold
All-Cause Mortality (participants affected / at risk) | 146/903 | 135/901
Serious Adverse Events (participants affected / at risk) | 206/908 | 197/906
Other Adverse Events (participants affected / at risk) | 184/908 | 164/906
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Tranfusion Threshold (N=908) | Low Transfusion Threshold (N=906)
Hemolysis (Blood and lymphatic system disorders) | 1 | 0
Adrenal Insufficiency (Endocrine disorders) | 2 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Bell's stage > 2 Necrotizing Enterocolitis (NEC) (Gastrointestinal disorders) | 58 | 62
Bowel Obstruction (Gastrointestinal disorders) | 1 | 2
Esophageal Perforation (Gastrointestinal disorders) | 0 | 2
Ischemic Bowel (Gastrointestinal disorders) | 0 | 1
Spontaneous Intestinal Perforation (Gastrointestinal disorders) | 29 | 38
Severe Hemorrhage (General disorders) | 5 | 2
Nosocomial Sepsis up to 24 hours post-transfusion (Infections and infestations) | 31 | 22
Pneumonia (Infections and infestations) | 1 | 1
Sepsis Bacterial (Infections and infestations) | 3 | 0
Sepsis Fungal (Infections and infestations) | 0 | 3
Sepsis Viral (Infections and infestations) | 0 | 2
Severe Cellulitis (Infections and infestations) | 1 | 0
Hyperkalemia -- non-hemolyzed specimen, up to 24 hours post-transfusion (Metabolism and nutrition disorders) | 10 | 16
Seizures (Nervous system disorders) | 2 | 1
Renal Failure (Renal and urinary disorders) | 4 | 2
Persistent Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary Air Leaks (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 13 | 9
Respiratory Deterioration up to 24 hours post-transfusion (Respiratory, thoracic and mediastinal disorders) | 93 | 85
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Severe Hypotension (Vascular disorders) | 1 | 1
Thrombosis (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 0.05% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High Tranfusion Threshold (N=908) | Low Transfusion Threshold (N=906)
Hyperkalemia -- non-hemolyzed specimen, up to 24 hours post-transfusion (Metabolism and nutrition disorders) | 58 | 40
Respiratory Deterioration up to 24 hours post-transfusion (Respiratory, thoracic and mediastinal disorders) | 147 | 146

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators must adhere to the Neonatal Research Network Publication Policies

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-07): https://cdn.clinicaltrials.gov/large-docs/05/NCT01702805/Prot_SAP_000.pdf